CLINICAL TRIAL: NCT00002842
Title: Hepatic Resection Followed by Concurrent Adjuvant Portal Vein Infusion of Fluorodeoxyuridine and Systemic 5-Fluorouracil and Folinic Acid for Metastatic Colorectal Carcinoma
Brief Title: Liver Resection and Floxuridine Plus Fluorouracil and Leucovorin in Treating Patients With Liver Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94080; P30CA033572 (NIH); CHNMC-IRB-94080; NCI-V96-1031; CDR0000065077 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Fluorouracil; Leucovorin; Chemotherapy, Adjuvant

ARMS (1):
- Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin (Experimental): Patients receive floxuridine via portal vein infusion from days 1-14. Systemic chemotherapy consists of leucovorin calcium on days 8-14 and fluorouracil on days 9-13. Courses repeat every 4 weeks for a total of 12 weeks
  Interventions: Drug: floxuridine; Drug: fluorouracil; Drug: leucovorin calcium; Procedure: adjuvant therapy; Procedure: conventional surgery

INTERVENTIONS:
Drug: floxuridine — Starting dose of 0.2 mg/kg/day for 14 consecutive days.
Drug: fluorouracil — 300 mg/m2/day by intravenous bolus 24 hours apart for 5 consecutive days.
Drug: leucovorin calcium — 500 mg/m2/day by continuous intravenous infusion beginning 24 hours prior to the first dose of 5-FU and continuing until 12 hours following the last dose of 5-FU.
Procedure: adjuvant therapy — Chemotherapy given after hepatic resection
Procedure: conventional surgery — Hepatic resection

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving drugs in different ways may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of surgery followed by floxuridine plus systemic fluorouracil and leucovorin in treating patients with liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of hepatic resection followed by portal vein infusion of floxuridine plus systemic fluorouracil/leucovorin calcium in patients with metastatic colorectal cancer.
* Study the toxic effects of adjuvant chemotherapy following hepatic resection.
* Evaluate mRNA expression of enzymes that may be important to the cytotoxicity of fluoropyrimidines in tumor cells, including thymidylate synthase, ribonucleotide reductase, and folylglutamyl synthetase, by polymerase chain reaction and immunohistochemistry.

OUTLINE: Following resection of the liver and all extrahepatic colorectal cancer, patients receive floxuridine via portal vein infusion from days 1-14. Systemic chemotherapy consists of leucovorin calcium on days 8-14 and fluorouracil on days 9-13. Courses repeat every 4 weeks for a total of 12 weeks.

If biopsy-proven metastatic disease develops, treatment may be stopped at the investigator's discretion. Continuation of regional therapy should be considered for extrahepatic failure. No concurrent radiotherapy is permitted.

Patients are followed every 3 months for 3 years, then every 6 months for survival.

PROJECTED ACCRUAL: It is expected that 50 patients will be entered over approximately 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal carcinoma or radiologically confirmed colorectal carcinoma in a synchronous metastasis
* Intrahepatic metastases required

  * No more than 15 metastases involving no more than 60% of functioning liver
* No extrahepatic disease unless:

  * Resectable anastomotic or locally recurrent tumor
  * Resectable mesenteric lymph node involvement in patients undergoing initial resection of primary colorectal carcinoma
  * Disease extension from liver metastasis amenable to en bloc resection (e.g., diaphragm wall, kidney, abdominal wall)
* No biopsy-proven chronic active hepatitis

PATIENT CHARACTERISTICS:

Age:

* Physiologic 18 to 70

Performance status:

* Karnofsky 60%-100%

Hematopoietic:

* AGC at least 1,500
* Platelets at least 100,000

Hepatic:

* Bilirubin no greater than 2.0 mg/dL (unless reversibly obstructed by metastasis)

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No second malignancy within 5 years except adequately treated:

  * Nonmelanomatous skin cancer
  * In situ bladder cancer
  * In situ cervical cancer
  * No pregnant women

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior mitomycin or nitrosoureas allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the liver
* At least 3 weeks since radiotherapy and recovered
* Prior pelvic radiotherapy allowed
* No planned concurrent radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1994-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucille A. Leong, MD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin
Started | 49
Completed | 22
Not Completed | 27
Not completed — ineligible for surgical resection | 27

BASELINE CHARACTERISTICS:
Arm/Group | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 56 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: 2 Year Disease-free Survival .
Description: Estimated using the product-limit method of Kaplan and Meier. Disease free survival, defined as first documented evidence of treatment failure. Acceptable evidence includes: Anastomotic - positive cytology or biopsy; Abdominal, pelvic and retroperitoneal nodes - progressively enlarging node as evidenced by 2 CT scans separated by at least a 4 week interval, ureteral obstruction in the presence of a mass as documented on CT scan; Peritoneum - positive cytology or biopsy, progressively enlarged intraperitoneal solid mass as evidenced by 2 CT scans separated by at least 4 weeks; Ascites - positive cytology or biopsy; Liver - positive cytology or biopsy; Pelvic mass - positive cytology or biopsy, progressively enlarging intrapelvic solid mass as evidenced by 2 CT scans separated by at least 4 weeks; Abdominal wall - positive cytology or biopsy; Lung - positive cytology or biopsy or presence of multiple pulmonary nodules; Bone marrow - positive cytology, aspiration or biopsy.
Time Frame: 2 years after treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin
Number analyzed (Participants) | 22
percentage of participants | 9 [2 to 34]

ADVERSE EVENTS:
Time Frame: Adverse events occurring over a period of 7 years and 6 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin (N=22)
Diarrhea (Gastrointestinal disorders) | 2 (2)
AGC (Investigations) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Lymphopenia (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hepatic Resection/Portal Vein FUdr/Systemic 5-FU & Leucovorin (N=22)
Dysrhythmias (Cardiac disorders) | 2 (3)
Other Misc (General disorders) | 9 (14)
Pericardial (Cardiac disorders) | 1 (1)
Stomatitis (General disorders) | 7 (10)
Weight (Food Intake) (Metabolism and nutrition disorders) | 1 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 11 (26)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (8)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 20 (66)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (10)
Nausea (Gastrointestinal disorders) | 15 (31)
(Gastrointestinal disorders) | 3 (6)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (19)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 12 (20)
Fever (General disorders) | 3 (3)
Fever (no infection) (General disorders) | 7 (15)
Oedema NOS (General disorders) | 2 (7)
Pain (General disorders) | 2 (5)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
AGC (Investigations) | 5 (14)
Alanine aminotransferase increased (Investigations) | 11 (41)
Alkaline Phosphatase (Investigations) | 5 (18)
Alkaline phosphatase increased (Investigations) | 8 (26)
Aspartate aminotransferase increased (Investigations) | 12 (32)
Bilirubin (Investigations) | 1 (1)
Creatinine (Investigations) | 1 (2)
Creatinine increased (Investigations) | 1 (3)
HGB/HCT (Investigations) | 8 (32)
Hyperbilirubinemia (Investigations) | 2 (9)
INR increased (Investigations) | 5 (8)
Leukopenia (Investigations) | 10 (21)
Lymphopenia (Investigations) | 1 (3)
Neutrophil count decreased (Investigations) | 4 (7)
Platelet count decreased (Investigations) | 6 (12)
Platelets (Investigations) | 4 (17)
Prothrombin Time (Investigations) | 4 (6)
SGOT/SGT (Investigations) | 9 (39)
WBC (Investigations) | 7 (19)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (31)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (25)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (29)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cortical/State of Consciousness (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (4)
Motor Activity (Nervous system disorders) | 1 (1)
Peripheral Nervous System Sensory (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 5 (7)
Taste alteration (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (7)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mood (Psychiatric disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (6)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Local Skin Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (12)
Sweating (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes